CLINICAL TRIAL: NCT04115202
Title: Comparative Study of the Results of Anterior and Posterior Arthrodesis in Degenerative Lumbar Pathology
Acronym: ECALAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Pr Jérome Allain (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-A02319-44
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Lumbar Arthrodesis
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- posterior spinal approach group: Lumbar arthrodesis performed by a posterior spinal approach.
  Interventions: Procedure: lumbar arthrodesis
- anterior spinal approach group: Lumbar arthrodesis performed by a anterior spinal approach.
  Interventions: Procedure: lumbar arthrodesis

INTERVENTIONS:
Procedure: lumbar arthrodesis — two approaches anterior versus posterior, optimally by leaving physicians free to use them as they do daily without modifying their procedures

SUMMARY:
To compare the functional results through the improvement of the Oswestry medium-term score of the lumbar arthrodesis performed to treat patients with lumbago and/or lumbar-radicular pain due to degenerative lesions of the lumbar spine: degenerative disc disease, osteoarthritis spondylolisthesis or adult dislocation scoliosis.

DETAILED DESCRIPTION:
Lower back pain is the leading cause of disability in France for adults under 45 years of age. It is also the leading cause of work stoppage and reported occupational illnesses. Thus, the degenerative pathologies of the lumbar spine can be at the origin of a severe handicap resistant to well-conducted medical treatment. This is particularly the case for degenerative disc disease, osteoarthritic spondylolisthesis and scoliotic dislocations in adults.

If lumbar arthrodesis is a recognised solution in the surgical treatment of degenerative diseases of the lumbar spine when they become disabling despite medical treatment, the choice of the operative technique and approach used to achieve it is more dependent of the training that the practitioner benefited from than the guidelines derived from published prospective comparative scientific studies comparing the results of different surgical solutions.

Our hypothesis is that the functional and radiographic results of anterior lumbar arthrodesis techniques by minimally invasive approach may differ from those of conventional posterolateral arthrodesis.

We propose to compare the results of these two surgical techniques within the orthopedic and neurosurgeon team of the Institut Parisien du Dos, mastering these two approaches optimally by leaving them free to use them as they do daily without modifying their procedures. This should allow us to judge, in a well-defined population, whether one of the two techniques is superior to the other when performed by surgeons who are experienced in this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring a lumbar arthrodesis to be carried out by one of the seven investigative surgeons of the Geoffroy Saint Hilaire Clinic IPAD study.
* At least 18 years old (no upper age limit).
* Patient with chronic lumbago or lumbar radiculopathy and resistant to a conservative medical treatment sufficiently carried out for at least 6 months, included alongside the usual analgesic, anti-inflammatory, infiltration and rehabilitation contraindications.
* Patient whose lumbar and/or radicular VAS is greater than or equal to 50 mm
* Patient whose Oswestry Index is greater than or equal to 40%
* Patient responding on one anatomical level* to one of the following diagnoses:

  * Spondylolisthesis or degenerative retrolisthesis or
  * single stage dislocation on scoliosis or
  * degenerative disc disease without true disc herniation, without deformity and instability reaching a single anatomical level
  * *single-stage pathology located between L1 and the sacrum (1 stage = 2 vertebrae and an intervertebral disc).
* Patient with health insurance or beneficiary of a social security scheme
* Patient having been informed of and having agreed to the use of their health data (non-opposition)

Exclusion Criteria:

* - Any situation that is a contraindication to either surgical approach. For example, for the anterior approach: morbid obesity, a history of multiple abdomen surgical procedures, aneurysm of the operated abdominal aorta making retroperitoneal dissection dangerous, severe arteritis with risk of mobilisation of aortoiliac atheromatous plaque, previous radiotherapy (radiation in the path of the approach).
* Contraindication to the strategy under study or an act of evaluation: for example contraindication to imagery provided (Pace maker for MRI).
* Pathology located in L1L2 which against indicates the previous conventional approaches (need to disinsert the diaphragm).
* Patient with proven osteoporosis: femoral T-score > -2 SD (measurement of the lumbar spine is not relevant because disturbed by osteoarthritic phenomena with vertebral osteo-condensation) and imposing a circumferential arthrodesis: anterior and posterior.
* Patient with excluded disc herniation: hernia that cannot be removed by anterior route (NB: A simple hernia is not a non-inclusion criterion).
* Association with the single-stage pathology another lumbar lesion imposing to extend the act of arthrodesis and/or decompression to one or more spinal stages.
* Any situation that could interfere with the follow-up of this study, i.e. psychological instability, personal situation hindering the follow-up of the study).
* Patient having undergone lumbar surgery less than one year ago
* Protected patients: adults under guardianship, trusteeship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, lactating or parturient women
* Individuals hospitalised without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a degenerative lumbar pathology operated
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry medium-term score | 12 months
  The absolute value and improvement of the Oswestry score at 1 year compared to the preoperative score for the 2 populations of lumbar arthrodesis by anterior or posterior approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Geoffroy Saint Hilaire Clinic, Paris, IDF, France